CLINICAL TRIAL: NCT05003089
Title: A Randomized, Controlled, Partial-blind, Parallel-group Study Evaluating the Effect of Oral Administration of BAY 1834845 and BAY 1830839 Twice Daily for 7 Consecutive Days on Local and Systemic IRAK4 Pathway-related Challenges in Healthy Male Participants
Brief Title: A Trial to Learn How BAY1834845 and BAY1830839 Affect Inflammation When Taken by Mouth Twice a Day for 7 Days in a Row in Healthy Male Participants
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Bayer (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Basic Science
Other Study IDs: 21329; 2020-003138-18 (EudraCT Number)
Record Dates: First submitted 2021-07-16; First posted 2021-08-12 (Actual); Last update posted 2022-12-16 (Actual); Status verified 2022-12

CONDITIONS: Immune Mediated Inflammatory Diseases
MeSH Terms: interventions — zabedosertib; Prednisolone

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: Double blind for BAY1834845, BAY1830839 and placebo (participant and investigator) with unblinded active control (prednisolone), rater-blinded for skin reaction assessments (all 4 study interventions).
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- BAY1834845 arm (Experimental): BAY1834845 will be administered twice daily for 7 consecutive days (Days 1 - 7).
  Interventions: Drug: BAY1834845
- BAY1830839 arm (Experimental): BAY1830839 will be administered twice daily for 7 consecutive days (Days 1 - 7).
  Interventions: Drug: BAY1830839
- Prednisolone arm (Active Comparator): Prednisolone will be administered twice daily for 7 consecutive days (Days 1 - 7).
  Interventions: Drug: Prednisolone
- Placebo arm (Placebo Comparator): Placebo will be administered twice daily for 7 consecutive days (Days 1 - 7).
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: BAY1834845 — Tablet, oral.
  Arms: BAY1834845 arm
Drug: BAY1830839 — Tablet, oral.
  Arms: BAY1830839 arm
Drug: Prednisolone — Tablet, oral.
  Arms: Prednisolone arm
Drug: Placebo — Tablet, oral.
  Arms: Placebo arm

SUMMARY:
The immune system helps protect the body from diseases. But, sometimes the immune system can be too sensitive and overreact to very small allergens, like dust and pet dander. This can cause skin conditions like dermatitis and eczema. People with these skin conditions have inflammation that can cause dry, red, and itchy skin. These symptoms often "flare up", meaning that the symptoms come back after being gone for some time.

Researchers are looking for a different way to treat people who have skin conditions caused by an overreaction of the immune system. Before a treatment is available to all patients, researchers study it in trials to better understand its safety and how well it works.

In this trial, the researchers will learn more about how BAY1834845 and BAY1830839 work and how safe they are in healthy male participants.

The trial will include about 72 healthy male participants who are between the ages of 18 and 55.

The researchers will use a computer program to randomly choose the treatment each participant will take. This will help make sure the treatments are chosen fairly. Researchers do this so that comparing the results of the treatments is accurate as possible. The participants will be randomly put into 1 of 4 groups. The participants will take their trial treatment 2 times a day for 7 days in a row.

* Group 1: BAY1834845 as tablets by mouth
* Group 2: BAY1830839 as tablets by mouth
* Group 3: A placebo as tablets by mouth
* Group 4: Prednisolone as tablets by mouth A placebo looks like a treatment but does not have any medicine in it. Prednisolone is a steroid treatment that is already available for doctors to prescribe to people with skin conditions caused by an overreaction of the immune system.

All the participants will also receive imiquimod applied as a cream to their back. All participants will also receive lipopolysaccharide as an intravenous infusion. Imiquimod and lipopolysaccharide will be used to cause irritation and inflammation of the skin and in the blood. The researchers want to see if treatment with BAY1834845 and BAY1830939 can then help reduce these symptoms of irritation and inflammation.

In this trial, the researchers will look at:

* the change in the amount of blood flow in the participants after imiquimod
* the change in how red the participants' skin is after imiquimod
* the change in the amount of inflammation applying the participants have after receiving lipopolysaccharide infusion

ELIGIBILITY:
Inclusion Criteria:

* Participant must be 18 to 55 years of age inclusive, at the time of signing the informed consent.
* Overtly healthy as determined by medical evaluation including medical and surgical history, physical examination, laboratory tests, ECG and vital signs.
* Participant has Fitzpatrick skin phototypes I (very fair), II (fair), or III (darker white skin).
* Body weight must be above 50 kg and body mass index (BMI) above or equal 18.5 and lower or equal 28 kg/m2 at the screening visit.
* Male.

Exclusion Criteria:

* Medical disorder, condition or history of such that would impair the participant's ability to take part in or complete this study in the opinion of the investigator
* A history of relevant diseases of vital organs, of the central nervous system including neuropsychiatric illness or other organs, previous syncope or autoimmune disease such as multiple sclerosis, inflammatory bowel disease, rheumatoid arthritis or other immune-inflammatory diseases.
* Unintended weight loss or gain of at least 5 kg in 4 weeks at screening.
* Any serious concomitant illness that anticipates the need of systemic medication interfering with the study medication.
* A history of trauma with likely damage to the spleen, surgery to spleen or congenital abnormalities of the spleen.
* Hemorrhagic diathesis (easy bruising, epistaxis, gastro-intestinal bleeding).
* History of known pulmonary embolism or known anti-phospholipid syndrome.
* Previous participation in a systemic (i.v./inhalative) lipopolysaccharide (LPS) challenge trial within one year before start of treatment.
* Diseases for which it can be assumed that the absorption, distribution, metabolism, elimination and effects of the study intervention(s) will not be normal (cholecystectomy permitted).
* Any infection requiring hospitalization, systemic antimicrobial therapy within 60 days, or as otherwise judged to be an opportunistic infection or clinically significant by the investigator, within the past 6 months prior to treatment period.
* Any active or ongoing chronic infectious disease including periodontitis with the exception of common viral or fungal skin infections such as plantar warts or athlete's foot.
* Febrile illness within 30 days before the start of the first study intervention.
* Medical history of sepsis, tuberculosis, increased frequency of infections, immunodeficiency diseases, with recent febrile diseases and anamnestic and/or laboratory signs of an impaired immune status or latent infections (hepatitis B, hepatitis C, and human immunodeficiency virus [HIV]).
* History of COVID-19 within 6 months prior to treatment period or in case of clinically relevant sequela of former COVID-19 (such as fatigue or exercise dyspnea)
* Contact with SARS-CoV-2- positive or COVID-19 patient within the last 2 weeks prior to SARS-CoV-2 viral PCR test (at visit 2).
* History of major surgery within 8 weeks prior to treatment period or scheduled (elective) surgery, planned hospitalization and surgical dental treatment within study and 4 weeks after final follow-up.
* History of or acute atopic dermatitis with active eczematous lesions, bronchial asthma or allergic rhino-conjunctivitis symptomatic during screening period.
* History of other concomitant skin conditions (chronic inflammatory dermatoses) that would interfere with the evaluation of the effect of the study medication on contact dermatitis.
* History of hypersensitivity to any of the components of the study interventions.
* History of malignant tumors (except treated basal cell carcinoma).
* Any clinical contraindications to treatment with steroids, such as uncontrolled hypertension, chronic liver disease (Child-Pugh scores B or C), latent diabetes mellitus, history of gastrointestinal bleeding.
* Use of topical and systemic drugs (prescription or over-the-counter [OTC]) within 30 days or within 5 half-lives (whichever is longer) before start of treatment.
* Use of other investigational drugs within 30 days or within 5 halflives (whichever is longer) of the investigational product before screening.
* Receipt of live or attenuated vaccine (with the exception of adenovirus-vectored SARS-CoV-2 vaccinations) 90 days before start of treatment.
* Vaccination completion (completion of 2nd vaccination shot if applicable) against SARS-CoV-2 or influenza vaccinations less than 15 days prior to first study drug administration. (Vaccines with a single-dose scheme: Receipt of vaccination < 29 days before the planned first administration of the study intervention).
* Phototherapy and extensive sun/ ultraviolet (UV) exposure within 4 weeks prior screening and throughout study.
* Clinically relevant findings in the ECG, blood pressure and pulse rate, which in the opinion of the investigator(s), may put the participant at risk because of his participation in the trial
* Clinically relevant findings in the physical examination, especially skin abnormalities in the application area.
* Clinically relevant deviations of the laboratory parameters from reference ranges at screening, ALT>1.1 x ULN, AST>1.2 x ULN, total bilirubin > ULN, CRP>5 mg/L (above ULN or clinical or laboratory signs of infection) or other clinically relevant laboratory abnormalities.
* Whole blood or red blood cell donation, or any blood loss > 500 mL within 3 months prior to screening or donation of plasma within 14 days prior to screening.

Ages: 18 Years to 55 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 51 (Actual)
Dates: Start 2021-06-28 (Actual); Primary Completion 2021-12-16 (Actual); Study Completion 2022-01-20 (Actual)

PRIMARY OUTCOMES:
Average change of perfusion/basal flow | Pre-challenge and at 24 hour / 48 hour / 72 hour after start of skin challenge
  The change from baseline will be averaged over the changes at 24 hour / 48 hour / 72 hour assessments
Average change of erythema score | Pre-challenge and at 24 hour / 48 hour / 72 hour after start of skin challenge
  The change from baseline will be averaged over the changes at 24 hour / 48 hour / 72 hour assessments. Erythema score will be measured by Antera 3D camera.
Average change in TNF-α | From pre-challenge up to 6 hour after the systemic challenge
Average change in IL-6 | From pre-challenge up to 6 hour after the systemic challenge

SECONDARY OUTCOMES:
Change of perfusion/basal flow | Pre-challenge and at 24 hour / 48 hour / 72 hour after start of skin challenge
Change of erythema score | Pre-challenge and at 24 hour / 48 hour / 72 hour after start of skin challenge
  Erythema score will be measured by Antera 3D camera.
Average change of Clinician Erythema Assessment (CEA) score | Pre-challenge and at 24 hour / 48 hour / 72 hour after first administration of skin challenge
  Clinician Erythema Assessment (CEA) scale:
  0 - Clear skin with no signs of erythema; 1 - Almost clear, slight redness; 2 - Mild erythema, defined redness; 3 - Moderate erythema, marked redness; 4 - Severe erythema, fiery redness.
Changes in cytokines cells of skin suction blisters | From baseline up to 72 hour after first administration of skin challenge
  Skin suction blisters will be induced on the tape stripping and/or treated skin areas, allowing the collection of blister exudate for cytokine cell analysis.
Changes in immune cells of skin suction blisters | From baseline up to 72 hour after first administration of skin challenge
  Skin suction blisters will be induced on the tape stripping and/or treated skin areas, allowing the collection of blister exudate for immune cell analysis.
Changes in immune cells of blood samples | From pre-challenge up to 24 hour after systemic challenge
Changes in C-reactive protein (CRP) of blood samples | From pre-challenge up to 24 hour after systemic challenge
Changes in Procalcitonin (PCT) of blood samples | From pre-challenge up to 24 hour after systemic challenge
Changes in other inflammation markers of blood samples | From pre-challenge up to 24 hour after systemic challenge
Changes in temperature | From pre-challenge to 0.5 hour / 1 hour / 2 hour / 4 hour / 6 hour and 8 hour after systemic challenge
Changes in pulse rate | From pre-challenge to 0.5 hour / 1 hour / 2 hour / 4 hour / 6 hour and 8 hour after systemic challenge
Changes in systolic blood pressure | From pre-challenge to 0.5 hour / 1 hour / 2 hour / 4 hour / 6 hour and 8 hour after systemic challenge
Changes in diastolic blood pressure | From pre-challenge to 0.5 hour / 1 hour / 2 hour / 4 hour / 6 hour and 8 hour after systemic challenge

CONTACTS AND LOCATIONS:
Locations (1):
- Center for Human Drug Research, Leiden, Netherlands

IPD SHARING:
Plan to Share IPD: No
Availability of this study's data will later be determined according to Bayer's commitment to the EFPIA/PhRMA "Principles for responsible clinical trial data sharing". This pertains to scope, timepoint and process of data access. As such, Bayer commits to sharing upon request from qualified researchers patient-level clinical trial data, study-level clinical trial data, and protocols from clinical trials in patients for medicines and indications approved in the US and EU as necessary for conducting legitimate research. This applies to data on new medicines and indications that have been approved by the EU and US regulatory agencies on or after January 01, 2014. Interested researchers can use www.clinicalstudydatarequest.com to request access to anonymized patient-level data and supporting documents from clinical studies to conduct research. Information on the Bayer criteria for listing studies and other relevant information is provided in the Study sponsors section of the portal.